CLINICAL TRIAL: NCT03231332
Title: Long Term Effects of H.Pylori Eradication on Microbiome and Adverse Events
Brief Title: Effects of H.Pylori Eradication on Microbiome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Latvia (Other)
Collaborators: Latvian Biomedical Research and Study Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.1.1/16/A/272
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Human Microbiome
Keywords: Helicobacter pylori; Eradication; Microbiome; ESBL; GIT

STUDY DESIGN:
Intervention Model Description: Comparison between intervention groups and the group without intervention will be made
Masking Description: Active treatment will be provided unmasked in the treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- H.pylori Eradication index (Experimental): Microbiome diversity detection in Participants Positive for H.pylori and undergoing Eradication therapy with Clarythromycin-containing eradication therapy
  Interventions: Other: Microbiome Diversity detection
- Control (No Intervention): Microbiome diversity detection in Participants Without H.pylori Eradication therapy
- H.pylori Eradication comparative (Active Comparator): Microbiome diversity detection in Participants Positive for H.pylori and undergoing Eradication therapy with high dose Amoxicillin and bismuth containing eradication therapy
  Interventions: Other: Microbiome Diversity detection

INTERVENTIONS:
Other: Microbiome Diversity detection — detection of microbiome composition and detection of specific mutations in genes conferring resistance to antibiotics
  Arms: H.pylori Eradication comparative; H.pylori Eradication index

SUMMARY:
The aim of this Project is, within the scope of industrial research, to evaluate the long term effects of H.pylori eradication on microbiome (gut microbiome, upper respiratory tract microbiome) and lasting adverse events. In addition, the project aims to evaluate its effects on abundance and prevalence of extended-spectrum beta-lactamases coding genes and develop cost effective ESBL screening test prototype.

DETAILED DESCRIPTION:
The current international guidelines and expert working groups are encouraging "search-and-treat" strategy for H.pylori to prevent gastric cancer1, 2. The highest yield of this approach is expected in countries with high incidence of gastric cancer and high prevalence of H.pylori infection. This approach will be further supported by the Maastricht V European guidelines (manuscript in preparation). The rationale for this approach is that 1-2% of the infected individuals are developing gastric cancer; the International Agency for Research on Cancer has classified H.pylori infection as Class I carcinogen3, 4. A study in Matsu island with high gastric cancer risk has suggested that gastric cancer incidence can be decreased by 25% by such strategy5; the limitations, however, include lack of the control group.

Three recent meta-analysis have confirmed the cost-effectiveness of such approach6-8; of course, those are based on the limited currently available data on potential risks caused by population-based strategy application.

In the countries which are expected to benefit from the strategy most this would mean offering eradication treatment to the majority of population, e.g. in Latvia this would require antibiotic treatment to 79% of population9, and would change the current status of low antibiotic consumption country to an average consumption country. This could potentially result in adverse consequences unrelated to H.pylori.

In a country with low H.pylori resistance to clarithromycin (such as Latvia), the recommended H.pylori 1st-line standard eradication regimen would consist of clarithromycin in combination to either amoxicillin or metronidazole, and a proton-pump inhibitor; the duration would be at least 10 days10. Areas with higher H.pylori resistance to clarithromycin would require more aggressive treatment modalities, e.g. by including levofloxacin to the regimen. The potential adverse events caused by such therapies to microbiome are insufficiently studied; the expert opinion that are developing guidelines is generally limited to the consideration that 1-2 week single-time antibiotic treatment would be a minor and fully reversible intervention upon microbiome since according to the available statistic in many countries the average antibiotic intake rates one or several treatments per year in a subject.

However, from the limited data available, there is a clear message that even one-week treatment with macrolides (clarithromycin, azithromycin) is increasing the resistance of macrolide-resistant S.pneumoniae in pharynx in healthy volunteers; this difference was statistically significant within a period of 180 days11.

Thus the aim of this project proposal is to evaluate the long term effects of H.pylori eradication on Gastro intestinal tract (GIT) microbiome, evaluate its effects on abundance and prevalence of extended-spectrum beta-lactamases (ESBL) coding genes and develop cost effective ESBL screening test prototype. To reach this goal during within the scope of this project fecal samples will be collected of patients that are undergoing the eradication therapy at two time points: before the start eradication and one year after the final treatment. In order to decrease the number of feces samples that patients shall have to acquire and standardize the sampling procedure, participants should explore the possibility to employ fecal occult blood test containers. Since there are no conclusively positive reports on employment of these devices in such analyses within the scope of this research participants shall also develop an appropriate DNA extraction methodology. Further, employing Next generation sequencing based analyses participants shall determine the microbial community composition within each sample and through comparison of data from each time point participants should be able to estimate the long term effects of eradication therapy. Following this analysis participants should perform the identification of ESBL repertoire within each sample and also evaluation their abundances abundance. Similarly as in the case of community analysis the comparison of both time points shall allow to estimate the effects of eradication therapy. Following the acquisition of the data participants shall outsource the creation of ESBL screening test prototype, which shall be based on employment micro-bead technology.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with established H.pylori infection
* Individuals in whom H.pylori eradication therapy is indicated according to the international or national recommendations
* Individuals who agree to undergo H.pylori eradication therapy

Exclusion Criteria:

* Severely sick patients
* Individuals in whom H.pylori eradication therapy is contra-indicated due to any reasons
* Individuals unable or unwilling to provide a sample for microbiome testing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-07-29 (Actual); Primary Completion 2019-10-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of various H.pylori eradication regimens upon the gut microbiome | 6-36 months between the initial and the follow-up sample
  Gut microbiome

SECONDARY OUTCOMES:
Effects of various H.pylori eradication regimens upon adverse events in short term | 21-28 days following the expected starting data of the treatmennt
  Telephone interview following eradication
Effectiveness of various H.pylori eradication regimens | 1-12 months following eradication therapy
  Effectiveness of H.pylori eradication will be evaluated by 13C urea breath test (UBT). Initially, 14 day clarythromycin-containing triple therapy will be compared to 14-day amoxicillin and bismuth containing therapy
Effects of various H.pylori eradication regimens upon the pharyngeal microbiome | 6-36 months between the initial and the follow-up sample
  Pharyngeal microbiome before and after H.pylori eradication will be compared
Effects of various H.pylori eradication regimens upon long-lasting adverse events | 6 months - 10 years following eradication
  Adverse evens like symptoms of gastro-esophageal reflux disease, obesity, functional bowel disease will be addressed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Latvia, Riga, Latvia

REFERENCES:
- [Background] Herrero R, Parsonnet J, Greenberg ER. Prevention of gastric cancer. JAMA. 2014 Sep 24;312(12):1197-8. doi: 10.1001/jama.2014.10498. No abstract available. PMID 25247512
- [Background] Schistosomes, liver flukes and Helicobacter pylori. IARC Monogr Eval Carcinog Risks Hum. 1994;61:1-241. No abstract available. PMID 7715068
- [Background] IARC, Monographs on the evaluation of carcinogenic risks to humans, volume 100. A review of carcinogen - Part B: biological agents. 2011, Lyon: International Agency for Research on Cancer.
- [Background] Lee YC, Chen TH, Chiu HM, Shun CT, Chiang H, Liu TY, Wu MS, Lin JT. The benefit of mass eradication of Helicobacter pylori infection: a community-based study of gastric cancer prevention. Gut. 2013 May;62(5):676-82. doi: 10.1136/gutjnl-2012-302240. Epub 2012 Jun 14. PMID 22698649
- [Background] Areia M, Carvalho R, Cadime AT, Rocha Goncalves F, Dinis-Ribeiro M. Screening for gastric cancer and surveillance of premalignant lesions: a systematic review of cost-effectiveness studies. Helicobacter. 2013 Oct;18(5):325-37. doi: 10.1111/hel.12050. Epub 2013 Apr 9. PMID 23566268
- [Background] Lansdorp-Vogelaar I, Sharp L. Cost-effectiveness of screening and treating Helicobacter pylori for gastric cancer prevention. Best Pract Res Clin Gastroenterol. 2013 Dec;27(6):933-47. doi: 10.1016/j.bpg.2013.09.005. Epub 2013 Sep 27. PMID 24182612
- [Background] Moayyedi, P., Feasibility and cost effectiveness of population-based H. pylori eradication, in In: IARC Helicobacter pylori Working Group. Helicobacter pylori Eradication as a Strategy for Preventing Gastric Cancer. Lyon, France: International Agency for Research on Cancer (IARC Working Group Reports, No. 8); pp. 174-180
- [Background] Leja M, Cine E, Rudzite D, Vilkoite I, Huttunen T, Daugule I, Rumba-Rozenfelde I, Pimanov S, Liepniece-Karele I, Pahomova J, Purmalis K, Eglitis J, Pirags V, Dzerve V, Erglis A. Prevalence of Helicobacter pylori infection and atrophic gastritis in Latvia. Eur J Gastroenterol Hepatol. 2012 Dec;24(12):1410-7. doi: 10.1097/MEG.0b013e3283583ca5. PMID 23114744
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Malhotra-Kumar S, Lammens C, Coenen S, Van Herck K, Goossens H. Effect of azithromycin and clarithromycin therapy on pharyngeal carriage of macrolide-resistant streptococci in healthy volunteers: a randomised, double-blind, placebo-controlled study. Lancet. 2007 Feb 10;369(9560):482-90. doi: 10.1016/S0140-6736(07)60235-9. PMID 17292768
- [Result] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502